CLINICAL TRIAL: NCT03751358
Title: Magnetic Resonance Imaging Analysis of the Spread of Local Anesthetic Solution After Ultrasound-guided Erector Spinae Plane Blockade
Brief Title: ESP Volunteer LA Spread Controlled by MRI
Acronym: ESP-MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with MRI interpretation
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VINMECTC
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Regional Anesthesia
Keywords: ESP Thoracic; Spread Local anesthetic; Volunteer; Magnetic résonance imaging

STUDY DESIGN:
Intervention Model Description: Healthy volunteers accepting to have a Unilateral ESP block with an MRI after injection of Low volume of local anesthetic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unilateral Erector spinae plane block (Experimental): Thoracic unilateral Erector spinae plane block performed on the volunteer and analyse of the spread of local anesthetic by magnetic resonance imaging
  Interventions: Procedure: Unilateral Erector spinae plane block

INTERVENTIONS:
Procedure: Unilateral Erector spinae plane block — Magnetic résonance imaging
  Other Names: Injection of Low volume of local anesthetic

SUMMARY:
Background and Objectives: The Thoracic Erector Spinae Plane Blockade (ESPB) is a regional anesthesia technique recently described by Forero M in November 2016 , whereby local anesthetic (LA) is injected in the inter Fascial space between posteriorly the fascia of Erector Spinae Muscles (IFS-ESP) (the iliocostalis, longissimus, and spinalis muscles ) and anteriorly the inter-transverse ligament to achieve multi-metameric analgesia for thoracic or upper abdominal surgery.

Recent studies published showed controversies on the spread of the local anesthetic and also the clinical efficiency .

The clarification of mechanism of the paravertebral block is one example for the effectiveness of Magnetic Resonance imaging (MRI) in this context We therefore designed a prospective study in volunteers to examine the spread of LA via MRI investigation in correlation with the extent of somatic block after a standardized ultrasound (US) guided ESPB. Our study will study the spread at T4 or T5 level which is the level used for most of thoracic, cardiac and breast surgeries to determine if dye would spread anteriorly to the involve or igins of the ventral and dorsal branches of the spinal nerves.

Methods:

After ethical committee approval we will select 10 Healthy volunteers to perform Unilateral ESP single shot block with a very low dose of Local anesthetic (LA) (Ropivacaine 0.5% 1 mg/kg (Maximal dose recommended = 3 mg/kg ) mixed with 0,1ml gadolinium After injection an ultrasound image of the spread of the LA with an easy 3 Dimension will be acquired. 10 and 30 minutes after injection a MRI will be performed to analyze the ultrasound spread. An Evaluation of the extension of Sensory Blockade.

Patient will be kept under monitoring for 1,5 hours to assess any complication Sensory block will be assessed. At 1 week after the study day, all volunteers will undergo an investigation of the puncture sites to exclude puncture- related infection or hematoma.

Statistical analysis will be done The cranio-caudal spread of LA will be recorded (US + MRI) and described for each of the volunteers.

DETAILED DESCRIPTION:
Screening Visit Ten healthy volunteers aged between 18 and 45 year olds Will be enrolled in the study. Prior to inclusion in the study, we informed them about the nature, scope, and the procedures of the study and about the particular study-related risks.

Exclusion criteria were defined as follows:

* Anatomical abnormalities of the thoracic spine identified by physical examination.
* Body mass index ≥30 kg/m2
* Medical contra-indication for Conscious MRI

  * Claustrophobia
  * Metal implants (pacemaker and others)
* Known allergy or hypersensitivity against Ropivacaine or other amino-amide LAs
* Participation in another clinical study within the last 4 weeks prior to study
* Coagulopathies in the medical history
* Abnormalities in electrocardiography that are considered clinically relevant such as atrio-ventricular block or bradycardia After signing the informed consent, each volunteer will go under a general physical examination, including patient history and drawing of blood for the laboratory (red and white blood count, and standard blood coagulation parameters).

In addition, an electrocardiogram as well as determination of blood pressure and heart rate will be performed. when all inclusion criteria will be met, a bilateral cross-sectional ultrasound examination of the IFS-ESP at the thoracic 4 (T4) level will be performed to confirm a clear identification of the ultrasound landmarks

* Transverse process T4
* Anterior fascia of Erector Spinae Muscle
* Inter-transverse ligament The T4 level will be determined by counting the spinous processes from the seventh cervical vertebra (vertebra prominens) in a distal direction. The screening visit took place within 3 weeks before study.

Ultrasound-guided ESPB and MRI Investigation On the morning of study, the volunteers will be admitted to the clinical ward. A venous access will be inserted into an antecubital vein and standard cardiorespiratory monitoring will be established (electrocardiogram, noninvasive blood pressure, and Spo2).

The ultrasound-guided injection of LA inside the IFS-ESP will be performed under direct ultrasound guidance using a ultrasound system (Logic S8 GE healthcare ultrasound) with a 50-mm 7-15 MHz linear ultrasound transducer in a para sagittal lateral position with the scheduled blocking area above. The IFS-ESP will be visualized as our group is performing at the level of T4 transverse process (See Bellow Performance protocole in Images) The puncture area and the ultrasound probe will be prepared in a sterile manner, and a skin wheal was performed with 1 ml lidocaine 2%. Then, the puncture will be performed with a 21-G, 80-mm Facette tip needle and an injection line (Stimuplex D Plus, 0.71 Å~ 80 mm, 22G Å~ 3 ⅛ ," BBraun Melsungen AG) realizing an "in-plane" ultrasound guided technique. Once the tip of the needle was placed inside the IFS-ESP, 2 ml dextrose will be injected checking the caudal and cranial spread and also the "breathing sign". (See protocol of puncture bellow). After these safety tests performed : local anesthetic Ropivacaine 0.5% mixed with 0,1ml gadolinium will be injected as follow:

* Patient 40 to 49 kg = 8 mL= 40 mg of ropivacaine
* Patient 50 to 59 kg = 10 mL = 50 mg of ropivacaine
* Patient 60 to 69 kg = 12 mL = 60 mg of ropivacaine
* Patient over 70 Kg = 15 mL = 75 mg of ropivacaine Maximum dose of Ropivacaine = 3 mg/kg (International recommendations and manufacturer recommendation) After the injection of LA a manual 3D acquisition will be done ( GE easy 3D Software) will do recorded to visualize the spread of LA inside the IFS-ESP, then an MRI will be performed 10 minutes and 30 minutes after injection using a 3-Tesla unit, long spine coil, covering the whole spine. T2-weighted sequences will be performed in sagittal and coronal planes. Axial T2-weighted sequences with fat suppression will be added in the region of the fluid accumulation. Axial T1-weighted sequences in this region will be performed to identify or exclude hemorrhagic components. Slice thickness will be 3 mm. During MRI investigation, the volunteers will be monitored via the MRI Bluetooth monitoring system (Spo2 , electrocardiogram). The distribution pattern of LA inside the IFS-ESP will be evaluated by analyses of the T2-weighted, fluid-sensitive images. Starting at the T4 puncture level, the axial T2-weighted sequences will be analyzed in a cranial and caudal direction to evaluate the cranio-caudal spread of LA. Any distribution of LA outside the IFS-ESP : ventral to the inter-transverse ligament, epidural, paravertebral prevertebral, and contralateral) will be analyzed. All images will be investigated by the same radiologist Evaluation of Sensory Blockade Sensory block will be assessed by pinprick testing with 22-G short bevel needles in comparison with the contralateral dermatomes. The blocked area will be tested from the T1 dermatome at the anterior axillary line and at the parasternal space in a cranial and then in a caudal direction. If required, the C2-5 dermatomes will be tested at the neck. Each individual dermatome on the blocked side will be compared with the contralateral side. All assessments will be performed by one investigator. Assessments will be quantified with the following scale
* 0 =full feeling)
* 1 = reduced
* 2 = No feeling

Sensory scores will be evaluated at the following time points:

* Prior block
* 30 min after block before second MRI investigation
* 60 min after block
* 120 min after block
* 24 h after the block to check the full recovery Successful blockade in a specific dermatome will be defined when pinprick testing will be positive value = 2. Onset and duration of ESPB will be not evaluated, as this study is designed to investigate the spread of LA within the ESPB. The expansion of the ESPB will be investigated meticulously.

Observation after Injection of LA Inside the IFS-ESP The volunteers will be observed and monitored (Spo2, electrocardiogram, and noninvasive blood pressure) 3 h after performance of ESPB and discharged after that time. A dedicated study emergency telephone number will be provided in cases of any medical problems.

Management of Side Effects Decrease in heart rate and blood pressure ≥30% from initial values will be treated with 0.01 mg/kg glycorpyrrolate and repetitive doses of 2 mg etilefrine, respectively.

Any sign of toxicity by IV injection = LAST protocol with intra-lipid 20% and keep in closed observation for 12 hours (ASRA recommendation) Follow-up Investigation At 1 week after the study day, all volunteers will undergo an investigation of the puncture sites to exclude puncture- related infection or hematoma.

Statistical Analysis The cranio-caudal spread of LA will be recorded and described for each of the volunteers. Due to not-normally distributed nature of the data, we will use a one-tailed Wilcoxon test to compare the cranial versus the caudal spread of LA at the same side. Pearson correlation coefficient will be used to correlate the spread of LA with the sensory distribution of ESPB Data will be presented as median (interquartile range). A P < 0.05 will be considered as statistically significant. SPSS 17.0.1 will be used as statistical software (IBM Inc., Armonk, NY).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18 and 45 year old

Exclusion Criteria:

* Refusal of the volunteer
* Anatomical abnormalities of the thoracic spine identified by physical examination.
* Body mass index ≥30 kg/m2
* Medical contra-indication for Conscious MRI
* Claustrophobia
* Metal implants (pacemaker and others)
* Known allergy or hypersensitivity against Ropivacaine or other amino-amide LAs
* Participation in another clinical study within the last 4 weeks prior to study
* Coagulopathies in the medical history
* Abnormalities in electrocardiography that are considered clinically relevant such as atrio-ventricular block or bradycardia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Magnetic resonnance Imaging spread | 40 minutes after injection
  spread of the local anesthetic
Sensory blockade evaluation | 4 hours after local anesthetic injection
  Pinprick testing from cervical dermatomes to T12 dermatome

CONTACTS AND LOCATIONS:
Overall Officials: Huyen Vu Xuan, MD, Study Chair — Vinmec Healthcare System
Locations (1):
- VinMec INternational hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Taketa Y, Irisawa Y, Fujitani T. Ultrasound-guided erector spinae plane block elicits sensory loss around the lateral, but not the parasternal, portion of the thorax. J Clin Anesth. 2018 Jun;47:84-85. doi: 10.1016/j.jclinane.2018.03.023. Epub 2018 Apr 6. No abstract available. PMID 29631112
- [Background] Schwartzmann A, Peng P, Maciel MA, Forero M. Mechanism of the erector spinae plane block: insights from a magnetic resonance imaging study. Can J Anaesth. 2018 Oct;65(10):1165-1166. doi: 10.1007/s12630-018-1187-y. Epub 2018 Aug 3. No abstract available. PMID 30076575
- [Background] Marhofer D, Marhofer P, Kettner SC, Fleischmann E, Prayer D, Schernthaner M, Lackner E, Willschke H, Schwetz P, Zeitlinger M. Magnetic resonance imaging analysis of the spread of local anesthetic solution after ultrasound-guided lateral thoracic paravertebral blockade: a volunteer study. Anesthesiology. 2013 May;118(5):1106-12. doi: 10.1097/ALN.0b013e318289465f. PMID 23442752
- [Background] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Gan TJ, Robinson SB, Oderda GM, Scranton R, Pepin J, Ramamoorthy S. Impact of postsurgical opioid use and ileus on economic outcomes in gastrointestinal surgeries. Curr Med Res Opin. 2015 Apr;31(4):677-86. doi: 10.1185/03007995.2015.1005833. Epub 2015 Feb 10. PMID 25586296